CLINICAL TRIAL: NCT01263899
Title: A Phase 2 Safety and Efficacy Study of SB1518 for the Treatment of Advanced Lymphoid Malignancies
Brief Title: A Safety and Efficacy Study of SB1518 for the Treatment of Advanced Lymphoid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: S*BIO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB1518-2010-005; NCT01263795 (obsolete NCT alias)
Record Dates: First submitted 2010-12-16; First posted 2010-12-21 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Hodgkin Lymphoma; Mantle Cell Lymphoma; Indolent Lymphoma
Keywords: Lymphoid malignancies; Hodgkin lymphoma; Mantle Cell Lymphoma; Indolent Lymphoma; SB1518
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Mantle-Cell | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB1518 (Experimental)
  Interventions: Drug: SB1518

INTERVENTIONS:
Drug: SB1518 — SB1518 taken orally daily for 28 consecutive days in a 28 day cycle.

SUMMARY:
This is a Phase 2 study to assess the efficacy of SB1518 in the treatment of patients with advanced lymphoid malignancies including Hodgkin Lymphoma, Mantle Cell Lymphoma and Indolent Lymphoma (follicular lymphoma, lymphoplasmacytic lymphoma, marginal zone lymphoma and small lymphocytic lymphoma).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented diagnosis of one of the following lymphoid malignancies:
* Hodgkin Lymphoma;
* Mantle Cell Lymphoma;
* Indolent Lymphoma (including follicular lymphoma, lymphoplasmacytic lymphoma, marginal zone lymphoma and small lymphocytic lymphoma);
* Patients must have received at least one prior treatment regimen; patients with Hodgkin Lymphoma must have received an autologous stem cell transplant, refused or been deemed ineligible for stem cell transplant;
* Able to understand and willing to sign the informed consent form.

Exclusion Criteria:

* Any histology other than Hodgkin Lymphoma, Mantle Cell Lymphoma or Indolent Lymphoma;
* History of or active Central Nervous System (CNS) malignancy;
* Active graft-versus-host disease (GVHD);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Assess overall tumor response of SB1518 by CT/FDG-PET scan and bone marrow biopsy as applicable as a measure of efficacy | Every even numbered cycle from baseline to 30 days after the last dose of study medication
  Outcome Measure - To assess the efficacy of SB1518 in the treatment of patients with advanced lymphoid malignancies including Hodgkin Lymphoma, Mantle Cell Lymphoma and Indolent Lymphoma (follicular lymphoma, lymphophasmacytic lymphoma, marginal zone lymphoma and small lymphocytic lymphoma).

SECONDARY OUTCOMES:
Assess durability of response | Every even numbered cycle from baseline to 30 days after the last dose of study medication
  To assess the durability of response following SB1518 treatment in patients with advanced lymphoid malignancies.
Assess number of patients with adverse events as a measure of safety and tolerability | Every even numbered cycle from baseline to 30 days after the last dose of study medication
  To assess the safety and tolerability of SB1518 administered orally once daily in patients with advanced lymphoid malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, MD, Principal Investigator — MD Anderson Cancer Center at University of Texas, Houston; Jonathan Friedberg, MD, Principal Investigator — University of Rochester James P. Wilmot Cancer Center; Peter Martin, MD, Principal Investigator — Weill Medical College of Cornell University; Julie Vose, MD, Principal Investigator — University of Nebraska; Richard Klasa, MD, Principal Investigator — British Columbia Cancer Center - Vancouver Centre
Locations (5):
- United States (4):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Weill Medical College of Cornell, New York, New York
  - University of Rochester James P. Wilmot Cancer Center, Rochester, New York
  - MD Anderson Cancer Canter, Houston, Texas
- University of British Columbia, Vancouver, British Columbia, Canada